CLINICAL TRIAL: NCT00128934
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of a Combination of Levonorgestrel and Ethinyl Estradiol in a Continuous Daily Regimen in Subjects With Premenstrual Dysphoric Disorder
Brief Title: Study Evaluating Combination of Levonorgestrel (LNG) and Ethinyl Estradiol (EE) in Premenstrual Dysphoric Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0858A4-316; NCT00278720 (obsolete NCT alias)
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Menstruation Disturbances; Premenstrual Syndrome
Keywords: Premenstrual Syndrome (PMS); Hormone Therapy
MeSH Terms: conditions — Menstruation Disturbances; Premenstrual Syndrome | interventions — Ethinyl Estradiol-Norgestrel Combination

INTERVENTIONS:
Drug: levonorgestrel/ethinyl estradiol

SUMMARY:
The purpose of this study is to determine whether levonorgestrel (LNG)/ethinyl estradiol (EE) is effective in treating the symptoms of severe premenstrual syndrome (PMS).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, women aged 18 to 49 years.
* History of severe PMS symptoms over the last year, as determined by the investigator.
* Regular 21 to 35 day menstrual cycle for 2 months prior to first study visit.

Exclusion Criteria:

* Major depressive disorder requiring antidepressant treatment or hospitalization within the last 3 years.
* Contraindication to combination oral contraceptives.
* Use of antidepressants/anxiolytics within 10 days of screening and for the duration of the study.

Other exclusions apply.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 744 (Estimated)
Dates: Start 2005-08; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Mean change in average Daily Record of Severity of Problems (DRSP) 21-item total daily score

SECONDARY OUTCOMES:
Change from baseline in DRSP 21-item daily score based on the 5 days with the highest DRSP scores in each "estimated" treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (75):
- United States (64):
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Carmichael, California
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - Lakewood, Colorado
  - Longmont, Colorado
  - Middletown, Connecticut
  - New Haven, Connecticut
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Adventure, Florida
  - Clearwater, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - South Bend, Indiana
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Glen Burnie, Maryland
  - Boston, Massachusetts
  - Pittsfield, Massachusetts
  - Springfield, Massachusetts
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Fayetteville, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Medford, Oregon
  - Philadelphia, Pennsylvania
  - Wexford, Pennsylvania
  - East Providence, Rhode Island
  - Greer, South Carolina
  - Hilton Head Island, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Conroe, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Sandy City, Utah
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Lakewood, Washington
  - Renton, Washington
- Canada (11):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Hull, Quebec
  - MontrÃ©al, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Shawinigan, Quebec
  - Sherbrooke, Quebec

REFERENCES:
- [Derived] Halbreich U, Freeman EW, Rapkin AJ, Cohen LS, Grubb GS, Bergeron R, Smith L, Mirkin S, Constantine GD. Continuous oral levonorgestrel/ethinyl estradiol for treating premenstrual dysphoric disorder. Contraception. 2012 Jan;85(1):19-27. doi: 10.1016/j.contraception.2011.05.008. Epub 2011 Jul 13. PMID 22067793